CLINICAL TRIAL: NCT00302159
Title: A Phase II Clinical Trial of the Histone Deacetylase Inhibitor Valproic Acid in Combination With Temodar and Radiation Therapy in Patients With High Grade Gliomas: Multi-Institutional Trial
Brief Title: Valproic Acid With Temozolomide and Radiation Therapy to Treat Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kevin Camphausen, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060112; 06-C-0112; NCT00313664 (obsolete NCT alias)
Record Dates: First submitted 2006-03-11; First posted 2006-03-13 (Estimated); Results first posted 2014-06-24 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-07

CONDITIONS: High Grade Gliomas; Brain Tumors
Keywords: Chemotherapy; Radiation; Brain Tumor; GBM; Radiosensitizer; Glioblastoma; Glioblastoma Multiforme
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma | interventions — Chemotherapy, Adjuvant; Temozolomide; Valproic Acid; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Valproic Acid (Experimental): Orally 25mg/kg/day twice a day concurrently with radiation therapy and temozolomide.
  Interventions: Procedure: adjuvant therapy; Drug: Temozolomide; Drug: Valproic Acid; Radiation: Radiation therapy

INTERVENTIONS:
Procedure: adjuvant therapy
Drug: Temozolomide — Orally 75mg/m^2 first day of radiation until completion. Restart 4 weeks post radiation.
  Other Names: Temodar
Drug: Valproic Acid — Orally 25mg/kg/day twice a day concurrently with radiation therapy and temozolomide.
  Other Names: Depakote
Radiation: Radiation therapy — External beam radiation Monday-Friday in 2 Gy fractions to 60 Gy total.

SUMMARY:
Background:

* Radiation therapy with temozolomide (an anti-cancer drug) is standard therapy for treating brain tumors called glioblastomas.
* The drug valproic acid, currently approved for treating seizures, has been shown in laboratory tests to increase the radiosensitivity of glioma cells.

Objectives:

-To determine the effectiveness of adding valproic acid to standard treatment with radiation therapy and temozolomide for treating glioblastoma.

Eligibility:

-Patients 18 years of age and older with glioblastoma multiforme who have not been previously treated with chemotherapy of radiation.

Design:

* This Phase II trial will enroll 41 patients.
* Patients will receive radiation therapy to the brain once a day, Monday through Friday, for 6 1/2 weeks.
* Patients will take temozolomide once a day by mouth, Monday through Friday, during the period of radiation treatment. Starting 4 weeks after radiation therapy, patients will take temozolomide once a day for 5 days every 28 days for a total of six cycles.
* Patients will receive valproic acid by mouth twice a day beginning 1 week prior to the first day of radiation therapy and continuing until the completion of chemotherapy and radiation therapy.
* Patients will have follow-up visits 1 month after completing therapy, then every 3 months for 2 years, and then every 6 months for 3 years. Follow-up includes a physical examination, blood tests and magnetic resonance imaging of the brain.

DETAILED DESCRIPTION:
BACKGROUND:

* Histone deacetylase inhibitors (HDACi) have recently been shown to enhance the radiosensitivity of glioma cells both in vitro and in vivo.
* Valproic acid has also recently been demonstrated to be a potent HDAC.
* Valproic acid has a long clinical history in patients with and without brain tumors and is known to cross the blood-brain barrier. However, the use of valproic acid in combination with temozolomide and radiotherapy for patients with high-grade gliomas has never been tested.

OBJECTIVES:

-The primary measure of efficacy will be progression free survival and overall survival.

ELIGIBILITY:

* Patients greater than 18 years old
* Diagnosis glioblastoma multiforme
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Patients who have not been previously treated with chemotherapy or radiation

DESIGN:

* This is a Phase II trial to determine the efficacy of valproic acid in combination with external beam radiation therapy and temozolomide in patients with high-grade gliomas.
* Patients will be treated with external beam radiation therapy in a standard manner with temozolomide given daily during the radiation. The valproic acid will be administered daily beginning one week prior to the first day of irradiation and continuing until the completion of chemoradiation.
* We anticipate that accrual to this trial of 41 patients will take approximately 1 year.

ELIGIBILITY:
* INCLUSION CRITERIA:

Histological diagnosis:

Pathologically confirmed glioblastoma multiforme.

Histologic diagnosis of glioblastoma multiforme (GBM) will have been established by biopsy or resection no more than 6 weeks prior to enrollment.

The patient is a candidate for definitive external beam radiotherapy.

Patients must be older than 18 years with a life expectancy greater than 8 weeks.

Patients should have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.

Patients must have a primary medical oncologist in the community who is willing to collaborate with the Radiation Oncology Branch (ROB) staff in the clinical management of the patient, specifically in the prescription of Temozolomide and toxicity monitoring in the adjuvant phase.

Laboratory functions:

Adequate bone marrow function defined as a peripheral absolute granulocyte count of greater than 1500/mm^3, hemoglobin greater than 10gm/dL, and platelet count greater than 100,000/mm^3.

Adequate liver function, defined as bilirubin and serum glutamic oxaloacetic transaminase (SGOT)/serum glutamic pyruvic transaminase (SGPT) less than 2 x the upper limit of normal.

Serum creatinine less than 1.5 mg/dl.

Serum albumin greater than 0.75 x normal.

All patients or their legal guardian must sign a document of informed consent indicating their understanding of the investigational nature and the risks of this study BEFORE any of the protocol related studies are performed (this does not include routine laboratory tests or imaging studies required to establish eligibility).

Subjects of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while they are being treated on this study.

EXCLUSION CRITERIA

Prior therapy:

Patients who have previously received valproic acid.

Patients who have previously received radiation therapy to the brain.

Patients who have received chemotherapy for the treatment of their high grade glioma or who are currently receiving other investigational chemotherapeutic agents.

Patients with a known history of disorders of urea metabolism.

Concurrent therapy:

The concurrent use of sulfamethoxazole, salicylates or naproxen is not allowed.

Patients with a history of or concurrent second malignancy other than non-melanoma skin cancer or cervical cancer less than 3 years since GBM diagnosis.

Pregnant or breast-feeding females are excluded because of the potential mutagenic effects on a developing fetus or newborn.

Clinically significant unrelated systemic illness which in the judgement of the Principal or Associate Investigator would compromise the patient's ability to tolerate this therapy or are likely to interfere with the study procedures or results, including but not limited to Insulin dependent diabetes.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-03; Primary Completion 2013-06 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Camphausen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Davis FG, McCarthy BJ, Freels S, Kupelian V, Bondy ML. The conditional probability of survival of patients with primary malignant brain tumors: surveillance, epidemiology, and end results (SEER) data. Cancer. 1999 Jan 15;85(2):485-91. PMID 10023719
- [Background] Loeffler JS, Alexander E 3rd, Shea WM, Wen PY, Fine HA, Kooy HM, Black PM. Radiosurgery as part of the initial management of patients with malignant gliomas. J Clin Oncol. 1992 Sep;10(9):1379-85. doi: 10.1200/JCO.1992.10.9.1379. PMID 1325539
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-C-0112.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Valproic Acid: adjuvant therapy
  Temozolomide Orally 75mg/m^2 first day of radiation until completion. Restart 4 weeks post radiation.
  Valproic Acid Orally 25mg/kg/day twice a day concurrently with radiation therapy and temozolomide.
  Radiation therapy External beam radiation Monday-Friday in 2 Gy fractions to 60 Gy total.
Period: Overall Study
Arm/Group | Valproic Acid
Started | 43
Completed | 41
Not Completed | 2
Not completed — pt declined before treatment started | 1
Not completed — pt started Avastin | 1

BASELINE CHARACTERISTICS:
Arm/Group | Valproic Acid
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.88 (11.33)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 35
  More than one race | 0
  Unknown or Not Reported | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival.
Description: Progression free survival is the interval from initiation of treatment on protocol to symptomatic or radiographic progression. Progressive disease is a >25% increase in contrast enhancing tumor volume documented at the initiation of treatment on protocol.
Time Frame: up to 51 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Valproic Acid
Number analyzed (Participants) | 43
months | 10.5 [7 to 51]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 6 years, 7 months and 27 days
Measure: Number; unit: participants
Arm/Group | Valproic Acid
Number analyzed (Participants) | 43
participants | 43

3. Primary Outcome: Percentage of Participants With Progression Free Survival at 6, 12, and 24 Months
Description: Percentage of participants who were progression free by 6, 12, or 24 months. Progressive disease is a >25% increase in contrast enhancing tumor volume documented at the initiation of treatment on protocol.
Time Frame: 6, 12, and 24 months
Measure: Number; unit: percentage of participants
Groups:
- Valproic Acid: Orally 25mg/kg/day twice a day concurrently with radiation therapy and temozolomide.
  adjuvant therapy
  Temozolomide: Orally 75mg/m^2 first day of radiation until completion. Restart 4 weeks post radiation.
  Valproic Acid: Orally 25mg/kg/day twice a day concurrently with radiation therapy and temozolomide.
  Radiation therapy: External beam radiation Monday-Friday in 2 Gy fractions to 60 Gy total.
Arm/Group | Valproic Acid
Number analyzed (Participants) | 43
percentage of participants
  6 months | 70
  12 months | 43
  24 months | 38

4. Primary Outcome: Number of Participants With Best Response
Description: Best response recorded from the start of treatment until disease progression/recurrence. Complete response is complete resolution of all contrast enhancing tumor documented at initiation of treatment on protocol, with no appearance of new lesions. Partial response is a >50% reduction in the contrast enhancing tumor volume documented at the initiation of treatment on protocol. Minor response is a >25%, but <50% reduction in the contrast enhancing tumor volume documented at the initiation of treatment on protocol. Stable disease is a change in tumor size less than MR but not demonstrating progressive disease. Progressive disease is a >25% increase in contrast enhancing tumor volume documented at the initiation of treatment on protocol. Not evaluable means the participant cannot be evaluated (e.g., quality of scan).
Time Frame: up to 63.8 months
Measure: Number; unit: participants
Arm/Group | Valproic Acid
Number analyzed (Participants) | 43
participants
  Complete Response | 0
  Partial Response | 0
  Minor Response | 0
  Stable Disease | 27
  Progressive Disease | 7
  Not Evaluable | 9

5. Primary Outcome: Median Overall Survival
Description: Survival is the interval from the initiation of treatment on protocol to date of death.
Time Frame: up to 63.8 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Valproic Acid
Number analyzed (Participants) | 43
months | 29.6 [21 to 63.8]

6. Primary Outcome: Percentage of Participants With Overall Survival at 6, 12, and 24 Months
Description: Percentage of participants who were alive at 6, 12, and 24 months.
Time Frame: 6, 12, and 24 months
Measure: Number; unit: percentage of participants
Arm/Group | Valproic Acid
Number analyzed (Participants) | 43
percentage of participants
  6 months | 97
  12 months | 86
  24 months | 56

ADVERSE EVENTS:
Arm/Group | Valproic Acid
Serious Adverse Events (participants affected / at risk) | 17/43
Other Adverse Events (participants affected / at risk) | 39/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valproic Acid (N=43)
Amylase (Metabolism and nutrition disorders) | 1 (1)
Ataxia (incoordination) (Nervous system disorders) | 3 (3)
Confusion (Nervous system disorders) | 2 (2)
Death not associated with CTCAE term::Disease progression NOS (General disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1)
Hemorrhage, CNS (Nervous system disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Infection - Other (Specify, pneumonia) (Infections and infestations) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Metabolic/Laboratory - Other (Specify, high ammonia) (Metabolism and nutrition disorders) | 1 (1)
Mood alteration::Agitation (Nervous system disorders) | 2 (2)
Neuropathy: motor (Nervous system disorders) | 3 (3)
Pain::Head/headache (Nervous system disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 2 (3)
Pulmonary/Upper Respiratory - Other (Specify, PE) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seizure (Nervous system disorders) | 4 (4)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 2 (2)
Vision-blurred vision (Eye disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Valproic Acid (N=43)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 15 (19)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 6 (7)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 27 (41)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (2)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 4 (4)
Amylase (Metabolism and nutrition disorders) | 6 (9)
Anorexia (Gastrointestinal disorders) | 6 (7)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (incoordination) (Nervous system disorders) | 10 (15)
Auditory/Ear - Other (Specify, decreased hearing) (Ear and labyrinth disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 7 (10)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 5 (5)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 4 (6)
Cardiac General - Other (Specify, systolic ejection murmur noted) (Cardiac disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Confusion (Nervous system disorders) | 16 (19)
Constipation (Gastrointestinal disorders) | 17 (19)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Creatinine (Metabolism and nutrition disorders) | 5 (6)
Cushingoid appearance (e.g., moon face, buffalo hump, centripetal obesity, cutaneous striae) (Endocrine disorders) | 2 (2)
Dehydration (Gastrointestinal disorders) | 2 (2)
Dermatology/Skin - Other (Specify, cyst R axilla) (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Dizziness (Nervous system disorders) | 5 (7)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 2 (2)
Edema: head and neck (Blood and lymphatic system disorders) | 4 (4)
Edema: limb (Blood and lymphatic system disorders) | 4 (5)
Encephalopathy (Nervous system disorders) | 2 (2)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 2 (3)
Extremity-upper (function) (Musculoskeletal and connective tissue disorders) | 1 (1)
Eyelid dysfunction (Eye disorders) | 1 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 25 (34)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - Other (Specify, GERD) (Gastrointestinal disorders) | 1 (1)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (8)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 23 (23)
Hearing: patients without baseline audiogram and not enrolled in a monitoring program (Ear and labyrinth disorders) | 2 (2)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 13 (23)
Hemorrhage, GI::Anus (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GU::Vagina (Reproductive system and breast disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 1 (1)
Incontinence, urinary (Renal and urinary disorders) | 2 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils::Conjunctiva (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Middle ear (otitis media) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Skin (cellulitis) (Infections and infestations) | 2 (2)
Infection with unknown ANC::Bronchus (Infections and infestations) | 1 (1)
Infection with unknown ANC::Paranasal (Infections and infestations) | 1 (1)
Infection with unknown ANC::Skin (cellulites) (Infections and infestations) | 1 (1)
Insomnia (General disorders) | 7 (7)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 14 (42)
Lipase (Metabolism and nutrition disorders) | 6 (10)
Lymphatics - Other (Specify) (Blood and lymphatic system disorders) | 2 (3) — L facial edema; Tonsillar edema; Mobile node L axilla
Lymphopenia (Blood and lymphatic system disorders) | 27 (79)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 15 (18)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 3 (3)
Memory impairment (Nervous system disorders) | 8 (8)
Mental status (Nervous system disorders) | 1 (1)
Metabolic/Laboratory - Other (Specify) (Metabolism and nutrition disorders) | 4 (6) — Elevated LD; Hypokalemia; Low protein; Phosphorus elevated
Mood alteration::Agitation (Nervous system disorders) | 6 (7)
Mood alteration::Anxiety (Nervous system disorders) | 5 (7)
Mood alteration::Depression (Nervous system disorders) | 4 (4)
Mood alteration::Euphoria (Nervous system disorders) | 1 (2)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 2 (2)
Mucositis/stomatitis (functional/symptomatic)::Oral cavity (Gastrointestinal disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy)::Extremity-upper (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscle weakness, generalized or specific area (not due to neuropathy)::Facial (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy)::Left-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy)::Right-sided (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal/Soft Tissue - Other (Specify, ® rotator cuff injury) (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 23 (30)
Neurology - Other (Specify) (Nervous system disorders) | 5 (5) — Dizziness; Hyperreflexivity; Decreased affect; Decreased attention span; Pronator drift
Neuropathy: cranial::CN II Vision (Nervous system disorders) | 1 (1)
Neuropathy: cranial::CN V Motor-jaw muscles; Sensory-facial (Nervous system disorders) | 2 (2)
Neuropathy: cranial::CN VII Motor-face; Sensory-taste (Nervous system disorders) | 1 (1)
Neuropathy: cranial::CN VIII Hearing and balance (Nervous system disorders) | 1 (2)
Neuropathy: motor (Nervous system disorders) | 11 (12)
Neuropathy: sensory (Nervous system disorders) | 6 (10)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 8 (16)
Nystagmus (Eye disorders) | 2 (2)
Ocular/Visual - Other (Specify) (Eye disorders) | 3 (3) — "Seeing shapes" in cloth; Eye irritation; Problems seeing bright lights
Otitis, middle ear (non-infectious) (Ear and labyrinth disorders) | 1 (2)
Pain - Other (Specify,jaw; right shoulder; whole body) (General disorders) | 2 (3)
Pain::Abdomen NOS (Gastrointestinal disorders) | 3 (4)
Pain::Back (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain::Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain::Dental/teeth/peridontal (Gastrointestinal disorders) | 1 (1)
Pain::Esophagus (Gastrointestinal disorders) | 1 (1)
Pain::External ear (Ear and labyrinth disorders) | 1 (1)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain::Head/headache (Nervous system disorders) | 14 (20)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain::Pain NOS (General disorders) | 1 (2)
Pain::Scalp (Skin and subcutaneous tissue disorders) | 2 (2)
Pain::Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pancreatitis (Hepatobiliary disorders) | 2 (2)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Blood and lymphatic system disorders) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (3)
Platelets (Blood and lymphatic system disorders) | 27 (63)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 14 (26)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (2)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 2 (2)
Pulmonary/Upper Respiratory - Other (Specify, pulomonary embolism) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pyramidal tract dysfunction (Nervous system disorders) | 1 (1) — (e.g., increased tone, hyperreflexia, positive Babinski, decreased fine motor coordination)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 (5)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 2 (3)
Rash: dermatitis associated with radiation::Chemoradiation (Skin and subcutaneous tissue disorders) | 4 (4)
Rash: dermatitis associated with radiation::Radiation (Skin and subcutaneous tissue disorders) | 5 (6)
Seizure (Nervous system disorders) | 11 (18)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 11 (16)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 11 (20)
Somnolence/depressed level of consciousness (Nervous system disorders) | 6 (6)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 4 (5)
Supraventricular and nodal arrhythmia::Sinus tachycardia (Cardiac disorders) | 1 (1)
Sweating (diaphoresis) (General disorders) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 4 (4)
Tremor (Nervous system disorders) | 4 (6)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 6 (9)
Vision-blurred vision (Eye disorders) | 4 (4)
Vision-flashing lights/floaters (Eye disorders) | 1 (1)
Vision-photophobia (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (8)
Watery eye (epiphora, tearing) (Eye disorders) | 2 (2)
Weight gain (General disorders) | 1 (1)
Weight loss (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No